CLINICAL TRIAL: NCT03127150
Title: Observational Study in Chyle Leak After Pancreatic Operation
Brief Title: Chyle Leak After Pancreatic Operation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZhejiangU05
Record Dates: First submitted 2017-04-04; First posted 2017-04-25 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
Keywords: Chylous leakage; Diagnostic criteria; Pancreas surgery; Therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CL group: Subjects who had CL after pancreatic operation will be observed.
- Observation group: Subjects without CL after pancreatic operation will be observed.

SUMMARY:
With the development of pancreatic surgery, the surgeon has put more emphasis on chylous fistula as the postoperative complications in recent years. The diagnostic criteria and treatment methods about chylous leakage have been developed and improved in clinical practice. However, there remains controversy about the high risk factors and efficient control measures during the perioperative period.

DETAILED DESCRIPTION:
Chylous fistula is one of the common complications after pancreatic operation, whose incidence is about 10%. The delayed diagnosis or wrong treatment in the perioperative period may lead to refractory chylous ascites, water-electrolyte imbalance, malnutrition, immune dysfunction, secondary infection and other complications. In the past, chylous fistula, as the postoperative complication, is common in abdominal aortic surgery, gynecological malignancies accompanied with posterior peritoneum lymphadenectomy and spinal surgery, etc. But chylous fistula after pancreatic operation did not attract enough attention. The comparative study or case analysis is lacked in relevant reports and there is no consensus on diagnostic criteria. In addition, once it occurs after pancreatic operation, the rehabilitation of patients will be affected, increasing the burden of hospitalization and even endangering the lives of patients due to the lack of diagnosis and treatment experience of specialists. The International Study Group of Pancreatic Surgery (ISGPS) proposed relevant definitions under the background of no unified diagnostic criteria of chylous fistula after pancreatic operation. But this definition still has some shortcomings; for example, it lacks the value of clinical guidance and research implementation. Moreover, how to take targeted preventive measures, choose the optimal treatment method and avoid complications, and whether there is a superior treatment method need to be further considered and investigated. Therefore, we performed this study, so as to better improve the relevant definition and provide guidance for the diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of CL after pancreatic operation
* Aged 18 or older
* Of either sex

Exclusion Criteria:

* No specific exclusion criteria will be applied to a participant as long as the participant is eligible for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed CL after pancreatic operation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Chylous fistula | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  The determine of chylous fistula follows the International Study Group on Pancreatic Fistulas (ISGPF) criteria.

SECONDARY OUTCOMES:
Extubation time | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  The time of removing the drainage tube
Hospital stays | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  the time during the operation to hospital discharge
Number of hospitalizations | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  Number of hospitalizations during the observational period
Mortality | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  Postoperative death in 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Bo Liang, phD, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No